CLINICAL TRIAL: NCT05056038
Title: The Comparison of Ultrasound-Guided Lateral and Posterior Quadratus Lumborum Block in The Pediatric Patients Undergoing Orchiopexy. A Double Blind Randomized Controlled Trial
Brief Title: Lateral Versus Posterior Quadratus Lumborum Block in The Pediatric Patients Undergoing Orchiopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozgecan Piril Zanbak, Attending Physician, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 90211
Record Dates: First submitted 2021-06-02; First posted 2021-09-24 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pain
Keywords: quadratus lumborum block; pediatric patient; orchiopexy; pain; regional anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Quadratus Lumborum Block (Active Comparator): After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both groups and the local anesthetic agent will be administrated with ultrasound at the anterolateral border of quadratus lumborum muscle with 18, 20 or 22 Gauge IV Cannula (Bıçakçılar Cooperation, Istanbul, Turkey) according to age and body weight.
  Interventions: Procedure: Lateral Quadratus Lumborum block
- Posterior Quadratus Lumborum Block (Active Comparator): After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both groups and the local anesthetic agent will be administrated with ultrasound at the posterior border of quadratus lumborum muscle with 18, 20 or 22 Gauge IV Cannula (Bıçakçılar Cooperation, Istanbul, Turkey) according to age and body weight.
  Interventions: Procedure: Posterior Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Lateral Quadratus Lumborum block — Local anesthetic may spread to the T6-L1 spinal nerves and paravertebral area by spreading through the lateral QLB to the transversus abdominis plane, and posteriorly via the anterior thoracolumbar fascia.
  Arms: Lateral Quadratus Lumborum Block
Procedure: Posterior Quadratus Lumborum Block — In posterior QLB, the local anesthetic can spread on the anterior and lateral cutaneous branches of T4-L1 spinal nerves by administration of the agent to the lateral interfascial triangle.
  Arms: Posterior Quadratus Lumborum Block

SUMMARY:
There is a complex innervation of the testis and spermatic canal, and many different regional analgesia methods can be used for pain occurring during and after undescended testicular surgery. Quadratus lumborum block (QLB) can be count as the one of the primary method to manage the pain.

In this study, our primary aim will be to compare the effects of lateral and posterior QLB application on perioperative and postoperative pain and analgesic use in pediatric patients who will undergo unilateral elective undescended testicular surgery. Our secondary aim will be to compare patient and family satisfaction and complications.

DETAILED DESCRIPTION:
American Society of Anesthesiologists Physical Status Classification System (ASA) class I-III, aged 6 month-12 years old children undergoing unilateral elective orchiopexy with general anesthesia will be recruited, after the informed consent will be obtained from the parents of the patients, in this triple blind randomized controlled trial.

After the premedication with ketamine and midazolam will be performed, the patient will be brought to the operation room. After the induction with thiopental 5mg/kg, fentanyl 1mcg/kg, rocuronium 0.6mg/kg, patients will be intubated. The maintenance of the anesthesia will be provided with sevoflurane.

Subsequently, before the surgery, the patients will be randomized and separated into 2 groups. The investigators will apply the lateral QLB to the first group and posterior QLB to the other group. 0.4 ml/kg %0.25 bupivacaine will be used as a local anesthetic agent in both group.

In the peroperative period, if the additional analgesia will necessary, remifentanyl 0.1mcg/kg/min will be started, and dosage will be adjusted according to heart rate and blood pressure. If the blood pressure or heart rate will increase more than 20% from the preoperative basal value will be defined as the need for the analgesia.

In the postoperative period, all cohort will be assessed by a blinded investigator at the 10,20,30th minutes, 1,2nd hours in the recovery room, 6th hour in the surgical ward, Face, Legs, Activity, Cry, Consolability Scale (FLACC) will be used for the pain evaluation. 16th and 24th hours will be monitored by the telephone visit from the parents, the pain will be evaluated with the Wong-Baker Faces Pain Rating Scale due to the same-day surgery concept.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Undergoing elective unilateral orchiopexy

Exclusion Criteria:

* Not giving a consent
* Regional anesthesia contraindications
* ASA physical status IV
* Need to postoperative ICU care
* Laparoscopic orchiopexy

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The Effect on Perioperative and Postoperative Pain | 24 hour
  The Face Legs Activity Cry Consobility (FLACC) Score will be used in hospital. The FLACC pain assessment score is evaluated out of 10 points. While a score of zero defined as no pain, 1-3 is mild pain, 4-6 is moderate pain, 7-10 is severe pain, respectively. If the score is 4 and above, additional analgesic administration will be planned. For the evaluation of the post-discharge, Wong Baker Pain score will be used. According to Wong Baker Score Pain will be evaluated based on six facial expressions between zero and ten points. If the score is four or more, additional analgesic administration will be planned.
Perioperative and Postoperative Total Analgesia Consumption | 24 hour
  The perioperative necessity of the additional analgesia was determined as the 20% increase of the heart rate and blood pressure values from the basal level and the dose of the remifentanyl was adjusted according to this protocol. The Face Legs Activity Cry Consobility (FLACC) Score will be used in hospital. The FLACC pain assessment score is evaluated out of 10 points. While a score of zero defined as no pain, 1-3 is mild pain, 4-6 is moderate pain, 7-10 is severe pain, respectively. If the score is 4 and above, additional analgesic administration will be planned. For the evaluation of the post-discharge, Wong Baker Pain score will be used. According to Wong Baker Score Pain will be evaluated based on six facial expressions between zero and ten points. If the score is four or more, additional analgesic administration will be planned.

SECONDARY OUTCOMES:
Parent satisfaction score | 24 hour
  At the postoperative 24th hour, the investigator will ask to the parents by telephone visit. Parent satisfaction score is defined as unsatisfied (1), partially satisfied (2), satisfied (3).
Complications | 24 hour
  The investigators will screen and record the complications such as nausea, vomiting, haematoma, solid organ injury, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Çiğdem Tütüncü, Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, McDonnell JG. Optimal point of injection: The quadratus lumborum type I and II blocks. Anaesthesia. 2013;68:4.
- [Background] Blanco R. Tap block under ultrasound guidance: the description of a "no pops" technique. Reg Anesth Pain Med. 2007;32:130.
- [Derived] Zanbak Mutlu OP, Kendigelen P, Tutuncu AC. Lateral versus posterior quadratus lumborum block in children undergoing open orchiopexy: a double-blind randomized clinical trial. Braz J Anesthesiol. 2025 Nov-Dec;75(6):844661. doi: 10.1016/j.bjane.2025.844661. Epub 2025 Jul 5. PMID 40623532